CLINICAL TRIAL: NCT02210572
Title: Effect of Prebiotics on Intestinal Gas Production, Microbiota and Digestive Symptoms
Brief Title: Effect of Prebiotics Versus Low FODMAPs Diet on Intestinal Microbiota and Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR(AG)296/2013/A-4/2014
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2014-08

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Intestinal microbiota; Intestinal gas; Dietary intervention; Low-FODMAPs diet; Prebiotics
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bimuno Galacto-oligosaccharide (Experimental): Dietary intervention
  Interventions: Dietary Supplement: Bimuno Galacto-oligosaccharide 1.37 g/d
- Low- FODMAPs diet (Placebo Comparator): Dietary intervention
  Interventions: Dietary Supplement: Low- FODMAPs diet

INTERVENTIONS:
Dietary Supplement: Bimuno Galacto-oligosaccharide 1.37 g/d — Prebiotic versus low-FODMAPs diet
  Arms: Bimuno Galacto-oligosaccharide
Dietary Supplement: Low- FODMAPs diet
  Arms: Low- FODMAPs diet

SUMMARY:
It has been shown that patients complaining of gas-related symptoms significantly improve on a diet low in fermentable residues. However, other studies suggest that some non-absorbable, fermentable meal products (prebiotics) that serve as substrate to colonic bacteria, produce beneficial effects to the host, including improvement of abdominal symptoms. The aim of the study is to compare the effects of a diet low in fermentable residues versus a diet suplemented with prebiotics on intestinal microbiota composition, microbiota activity (intestinal gas production) and digestive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Functional digestive disorder with flatulence
* Women and men between the ages of 18 and 80 years (bounds included at the inclusion visit).
* Normal body weight or with overweight (body mass index between 18.0 and 30.0 kg/m2 (bounds included)).
* Women of childbearing potential should be using or complying with one of the medically approved methods of contraception such as, but not exclusively, one of the following:

  1. Birth control pill
  2. Intra-uterine device (IUD)
  3. Double barrier methods (such as condoms and spermicide)
  4. Abstinence
* Willing to follow strict dietary instructions for the duration of the study
* Able to communicate well with the investigator and to comply with the requirements for the study.

Exclusion Criteria:

* Significant illness other than functional bowel disorders
* Disease/disorders which can interfere with the collection of the gas (hemorrhoids,..etc)
* Antecedents of digestive surgery, excluding appendicectomy
* Intake of antibiotics in the month (within 30 days) preceding the inclusion visit.
* Current use of any medications with potential central nervous system effects as judged by the investigator (including but not limited to antidepressants, anxiolytics, opiate pain medications)
* Taking drugs that might modify gastrointestinal function
* Change of dietary habits within the preceding 4 weeks (for instance start of a diet high in fiber) or planned change (For example to start a diet) during the period of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition | 28 days
  Effect of treatment on the response of microbiota to 3-day challenge diet

SECONDARY OUTCOMES:
Microbiota activity (intestinal gas production) | 28 days
  Intestinal gas evacuation on standardized diet
Digestive symptoms | 28 days
  Digestive sensations measured by scales

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, Principal Investigator — Vall d'Hebron Research Institute
Locations (1):
- Vall d'Hebron Research Institute, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Huaman JW, Mego M, Manichanh C, Canellas N, Canueto D, Segurola H, Jansana M, Malagelada C, Accarino A, Vulevic J, Tzortzis G, Gibson G, Saperas E, Guarner F, Azpiroz F. Effects of Prebiotics vs a Diet Low in FODMAPs in Patients With Functional Gut Disorders. Gastroenterology. 2018 Oct;155(4):1004-1007. doi: 10.1053/j.gastro.2018.06.045. Epub 2018 Jun 30. PMID 29964041